CLINICAL TRIAL: NCT05230732
Title: Neuromodulation of Inflammation and Endothelial Function to Treat Elderly Patients With Systolic Heart Failure
Brief Title: Neuromodulation of Inflammation and Endothelial Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14101; 5R21AG075639-02 (NIH)
Record Dates: First submitted 2022-01-10; First posted 2022-02-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Systolic Heart Failure
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental (Experimental): Active LLTS will be performed by use of a neuromodulation device with electrodes attached to the tragus of the ear. Stimulator will be applied continuously for 1 hour daily for 12 weeks.
  Interventions: Device: neuromodulation device
- Control arm (Sham Comparator): Sham LLTS will be performed by use of a neuromodulation device with electrodes attached to the ear lobule. Stimulator will be applied continuously for 1 hour daily for 12 weeks.
  Interventions: Device: SHAM

INTERVENTIONS:
Device: neuromodulation device — Active LLTS will be performed by use of a neuromodulation device with electrodes attached to the tragus of the ear. Stimulator will be applied continuously for 1 hour daily for 12 weeks
  Arms: Experimental
Device: SHAM — Sham LLTS will be performed by use of a neuromodulation device with electrodes attached to the ear lobule. Stimulator will be applied continuously for 1 hour daily for 12 weeks
  Arms: Control arm

SUMMARY:
Heart failure with reduced ejection fraction (HFrEF) is a major cause of mortality in United States. Aging is a major risk factor for adverse outcomes associated with HFrEF, with majority of the patient's over the age of 50, continuing to experience symptoms, reduced exercise capacity and poor quality of life. We have previously demonstrated that low level transcutaneous electrical stimulation of the vagus nerve at the tragus (LLTS) suppresses inflammation in patients with atrial fibrillation and diastolic dysfunction and improved endothelial dysfunction in patients with chronic heart failure. The overall objective of this proposal is to examine the effects of LLTS on heart failure symptoms, exercise capacity and quality of life in patients with HFrEF and simultaneously determine the impact of LLTS on the suppression of inflammation and improvement in endothelial function. Our specific aims include: 1. To examine the medium term effect of intermittent (1 hour daily for 3 months) LLTS on exercise capacity and quality of life, related to sham stimulation, in patients with HFrEF, 2. To determine the effects of medium-term LLTS on sympathovagal/autonomic balance (assessed by heart rate variability) and systemic inflammation in patients with HFrEF and 3. To determine the effects of medium-term LLTS on endothelial function in patients with HFrEF. The proposed proof-of-concept human studies will provide the basis for the design of further human studies using LLTS among larger populations with HFrEF. In light of the increasing number of elderly patients who continue to experience HFrEF symptoms, recognized is a key point of interest in this funding mechanism, and the suboptimal success of the currently available treatment options to ameliorate the problems mentioned above, an alternative novel approach such as LLTS has the potential to impact clinical practice and improve health outcomes among the large number of patients. It is anticipated that these investigations will contribute to a broader understanding of the role of autonomic imbalance, inflammation and endothelial dysfunction in the pathogenesis of HFrEF and how its inhibition can be used to provide therapeutic effects. Moreover, it is anticipated that a better understanding of how modulation of autonomic tone, inflammation and endothelial function affects one of the hallmarks of HFrEF will lead to the development of normal nonpharmacological and pharmacological approaches to treat this disease.

DETAILED DESCRIPTION:
Prospective randomized double-blind study of Lowlevel Tragus stimulation-LLTS vs. sham treatment.

We will require n=108 participants (54 in each group) to reach statistical significance and to account for potential drop-out (anticipated <5%, based on previous study in atrial fibrillation) from the study and 50 subjects below the age of 50 will be enrolled in the control group 2 for comparison purposes, for a total of 158 patients.

Aim 1:

Objective 1: measure the medium-term effects of LLTS on exercise capacity in subjects with HF - 6-minute walk distance (6MWD) will be performed at baseline and after 3 months of LLTS. Change in 6MWD from baseline to 3 months will be compared between experimental and sham groups. Duration of test: <10 minutes. A dedicated quite hallway exists in the translational geroscience laboratory which will enable performance of the test. Study will be performed by the research coordinator.

Objective 2: assess the effects of medium-term LLTS on quality of life in subjects with HF - quality of life will be determined using standard HF questionnaire (MLWHF score). This questionnaire will be administered at baseline and after 3 months. Duration of test: <15 minutes. Study will be administered by our research coordinator either on paper or tablet.

Aim2:

Objective 1: measure the effects of medium-term LLTS on sympathovagal balance in subjects with HF - Heart rate variability (HRV), a well-established, noninvasive measure of autonomic function, will be measured and analyzed via 10 min ECG using standard Labscribe and Kubios software. The amplitude and changes of the low (0.04-0.15Hz), high (0.15-0.4Hz) and the low frequency/high frequency ratio along with specific time domain variables (SDNN,SDANN,pNN50,rMSSD) will be determined to reflect autonomic imbalance.

Objective 2: assess the effects of medium-term LLTS stimulation on HF biomarkers, inflammation - using high sensitivity ELISA kits, NT-Pro BNP, sST2, Interleukins (6, 1), TNF-α, hsCRP will be assayed.

Aim 3:

Objective 1: assess the effects of medium-term LLTS on vascular endothelial function -Flow-mediated vasodilatation (FMD) will be used to assess %-change in brachial artery diameter upon the release of temporary 5-min blood flow occlusion to the extremity using ultrasonography (Phillips Affinity X70). This is a standard, validated technique to assess FMD. Average time to perform this study is ~20 minutes.

ELIGIBILITY:
Inclusion Criteria:

Systolic heart failure with EF < or equal to 50%.

Exclusion Criteria:

1. patients in overt congestive heart failure / recent acute myocardial infarction (< 4 weeks) or Unstable angina
2. Active malignancy
3. unilateral or bilateral vagotomy
4. pregnant patients
5. End stage liver disease
6. history of recurrent vasovagal syncope, Sick sinus syndrome with no pacemaker, 2nd or 3rd degree AV block.
7. Significant hypotension (Blood pressure < 90 mm Hg) secondary to autonomic dysfunction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
6MWD | Change in 6MWD after 12 weeks compared to baseline
  6 minute walk distance

SECONDARY OUTCOMES:
QoL | Change in QoL after 12 weeks compared to baseline
  Quality of life will be assessed using the Minnesota living with heart failure questionnaire

OTHER OUTCOMES:
FMD | Change in FMD after 12 weeks compared to baseline
  Flow mediated vasodilatation will be assessed using vascular ultrasound measuring brachial artery diameter change with standard 5 minute BP cuff occlusion test.
HRV | Change in HRV after 12 weeks compared to baseline
  heart rate variability
Inflammation | Change in inflammatory markers after 12 weeks compared to baseline
  Inflammatory cytokines will assayed at baseline and after 4 weeks of stimulation. Cytokines assayed : Il1B,IL-6,IL-17,TNF-a,TGF-b,CRP etc- expressed in pg/ml units).

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Dasari, MD, MPH, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No